CLINICAL TRIAL: NCT06015061
Title: Prediction and Evaluation of Anlotinib Treatment Response Using Contrast Enhanced Ultrasound in Patients With Pheochromocytoma or Paraganglioma
Brief Title: Prediction and Evaluation of Anlotinib Treatment Response Using Contrast Enhanced Ultrasound PPGL Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 06086-04
Record Dates: First submitted 2023-05-22; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-03

CONDITIONS: Pheochromocytoma, Metastatic; Ultrasonography; Paraganglioma, Malignant; Pheochromocytoma Malignant
MeSH Terms: conditions — Pheochromocytoma; Neoplasm Metastasis; Paraganglioma, Extra-Adrenal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pheochromocytoma or Paraganglioma Patients with Anlotinib Treatment: to evaluate the efficiency of contrast enhanced ultrasound in assessing effectiveness of anlotinib in patients with locally advanced, metastatic, or unresectable pheochromocytoma or paraganglioma(PPGL).
  Interventions: Diagnostic Test: Contrast-enhanced ultrasound(CEUS)

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced ultrasound(CEUS) — CEUS is a quantitative kinetic imaging modality that can assess intravascular blood flow in PPGL tumors.

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor (TKI) targeting tumor angiogenesis and growth. The purpose of this study is to evaluate the efficiency of contrast enhanced ultrasound in assessing effectiveness of anlotinib in patients with locally advanced, metastatic, or unresectable pheochromocytoma or paraganglioma(PPGL).

DETAILED DESCRIPTION:
Contrast-enhanced ultrasound (CEUS) is a non-invasive and efficient imaging technique which can observe the blood flow at the tissue perfusion level with microbubble contrast agents and obtain information about tumor perfusion. There have been several studies demonstrating the utility of CEUS for early prediction of response to neoadjuvant chemotherapy in breast cancer, pancrearic cancer as well as lymphoma. However, few studies have reported the use of CEUS for the evaluation of therapeutic response in PPGL. What quantitative parameters of CEUS can early reflect the neovascular changes after treatment with anlotinib in patients with locally advanced, metastatic, or unresectable PPGL? The aim of our study is to evaluate the parameters for CEUS imaging and the therapeutic response of PPGL before and after anlotinib therapy and to determine the most useful CEUS response parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Provide written informed consent.
* Willing to return to enrolling institution for follow-up.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Life expectancy > 3 months.
* Patients diagnosis with pheochromocytoma or paraganglioma will received anlotinib treatment.
* Laboratory requirements:

  * Absolute granulocyte count (AGC) greater than 1.5 x 109/L;
  * Platelet count greater than 80 x 109/L;
  * Hemoglobin greater than 90g/L;
  * Serum bilirubin less than 1.5 x upper limit of normal (ULN);
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN;
  * Serum creatinine less than 1.5 x ULN or creatinine clearance (CCr)≥60ml/min;
  * Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).

Exclusion Criteria:

* Patients who are allergic to ultrasound contrast agents.
* Any of the following:Pregnant women,Nursing women,Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Patients who have previously used other anti-vascular targeted drugs, such as sunitinib, bevacizumab, endurance, etc.
* Chemotherapy/systemic therapy, radiotherapy, immunotherapy or surgery within 4 weeks prior to kinase inhibitor therapy.
* Patients with another primary malignancy within 5 years prior to starting study drug.

Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.).

* Patients with known untreated brain metastases are excluded. Patients having a history of brain metastasis that have been previously irradiated or resected greater than 2 months prior to enrollment and are clinically and radiographically stable will be considered for enrollment. Patients with brain metastases with symptoms or symptom control for less than 2 months.
* Active or uncontrolled intercurrent illness including, but not limited to

  * Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg);
  * Patients with uncontrolled myocardial ischemia or myocardial infarction, arrhythmia (including QTC≥480ms), and uncontrolled congestive heart failure，grade ≥2（New York Heart Association )
  * ongoing or active infection;
  * Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment;
  * Renal failure requires hemodialysis or peritoneal dialysis;
  * Have a history of immunodeficiency, including HIV or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  * Diabetes is poorly controlled (fasting blood glucose (FBG)> 10mmol/L);
  * Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein content is confirmed to be greater than 1.0 g;
  * Patients who have seizures and need treatment;
* Any of the following conditions =< 6 months prior to registration: Cerebrovascular accident (CVA) or transient ischemic attack (TIA); Serious or unstable cardiac arrhythmia; Pulmonary embolism, untreated deep venous thrombosis (DVT).

Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment.

* Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders.
* Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study.
* Regardless of the severity, patients with any signs of bleeding or medical history; within 4 weeks before enrollment, patients with any bleeding or bleeding event ≥ CTCAE grade 3, unhealed wounds, ulcers or fractures.
* Patients are using drugs that interact with Anlotinib.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: in patients with locally advanced, metastatic, or unresectable pheochromocytoma or paraganglioma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate if tumor uptake of contrast agent is predictive of response to anlotinib therapy measured by comparison of Peak Intensity (PI) at CEUS imaging prior to and after therapy. | Baseline and after 1-2 cycles(each cycle is 21 days)
  Before initiation of the therapy and during anlotinib therapy, patients would receive CEUS examination. The dynamic CEUS images of each lesion were analysed with the aid of time intensity curves (TICs) drawn by QLAB software (Philips Healthcare, Andover, MA). PI measurements will be compared to clinical measurement of response to treatment taking into consideration standard response criteria including radiological imaging, biochemical (catecholamine levels) response.
Evaluate if the time to peak (TTP) is predictive of response to anlotinib therapy measured by comparison of TTP at CEUS imaging prior to and after therapy. | Baseline and after 1-2 cycles(each cycle is 21days)
  Before initiation of the therapy and during anlotinib therapy, patients would receive CEUS examination. The dynamic CEUS images of each lesion were analysed with the aid of time intensity curves (TICs) drawn by QLAB software (Philips Healthcare, Andover, MA). TTP measurements will be compared to clinical measurement of response to treatment taking into consideration standard response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Anli Tong, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim Y, Kim SH, Song BJ, Kang BJ, Yim KI, Lee A, Nam Y. Early Prediction of Response to Neoadjuvant Chemotherapy Using Dynamic Contrast-Enhanced MRI and Ultrasound in Breast Cancer. Korean J Radiol. 2018 Jul-Aug;19(4):682-691. doi: 10.3348/kjr.2018.19.4.682. Epub 2018 Jun 14. PMID 29962874
- [Result] Zhang Q, Wu L, Yang D, Qiu Y, Yu L, Dong Y, Wang WP. Clinical application of dynamic contrast enhanced ultrasound in monitoring the treatment response of chemoradiotherapy of pancreatic ductal adenocarcinoma. Clin Hemorheol Microcirc. 2020;75(3):325-334. doi: 10.3233/CH-190786. PMID 31985457
- [Result] Xin L, Yan Z, Zhang X, Zang Y, Ding Z, Xue H, Zhao C. Parameters for Contrast-Enhanced Ultrasound (CEUS) of Enlarged Superficial Lymph Nodes for the Evaluation of Therapeutic Response in Lymphoma: A Preliminary Study. Med Sci Monit. 2017 Nov 15;23:5430-5438. doi: 10.12659/msm.907293. PMID 29138385